CLINICAL TRIAL: NCT00021749
Title: Phase I-II Multicenter Study of Genasense (Bcl-2 Antisense Oligonucleotide) in Patients With Advanced Chronic Lymphocytic Leukemia
Brief Title: Phase I/II Study of Genasense in Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genta Incorporated (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GL208; G3139; Bcl-2 Antisense; NCT00021190 (obsolete NCT alias)
Record Dates: First submitted 2001-08-03; First posted 2001-08-06 (Estimated); Last update posted 2009-11-13 (Estimated); Status verified 2009-11

CONDITIONS: Chronic Lymphocytic Leukemia; CLL
Keywords: CLL; Leukemia; Chronic; Cancer; Adult; Lymphocytic; Genasense; G3139; Genta; Bcl-2; Antisense; Oligonucleotide; oblimerson
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia; Bronchiolitis Obliterans Syndrome; Neoplasms | interventions — oblimersen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Oblimerson sodium, G3139

SUMMARY:
This non-randomized study will test the safety and effectiveness of Genasense in patients with CLL.

DETAILED DESCRIPTION:
This study is a two-part phase I-II study. Part 1 will determine the MTD of Genasense in patients with CLL. This dose will then be tested in a non-randomized, multi-center, Phase II sequential clinical trial of Genasense used alone for treatment of patients with advanced CLL.

Pharmacokinetics of Genasense and kinetics of Bcl-2 down regulation and re-expression in CLL cells will be followed in selected patients.

ELIGIBILITY:
* Any age
* Must have received at least one chemotherapy regimen that included fludarabine
* Measurable disease
* At least 3 weeks since biological therapy or radiation therapy for chronic lymphocytic leukemia
* No previous stem cell transplantation
* At least 3 weeks since surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2001-01; Primary Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - MD Anderson Cancer Center, Houston, Texas
  - San Antonio Cancer Institute, San Antonio, Texas

REFERENCES:
- [Result] O'Brien SM, Cunningham CC, Golenkov AK, Turkina AG, Novick SC, Rai KR. Phase I to II multicenter study of oblimersen sodium, a Bcl-2 antisense oligonucleotide, in patients with advanced chronic lymphocytic leukemia. J Clin Oncol. 2005 Oct 20;23(30):7697-702. doi: 10.1200/JCO.2005.02.4364. Epub 2005 Sep 26. PMID 16186597